CLINICAL TRIAL: NCT02713178
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy, Safety, and Pharmacokinetics of Femoral Nerve Block With EXPAREL for Postsurgical Analgesia in Subjects Undergoing Total Knee Arthroplasty
Brief Title: Efficacy, Safety, and Pharmacokinetics of Femoral Nerve Block With EXPAREL in Total Knee Arthroplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 402-C-326
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Results first posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- EXPAREL 133 mg (Active Comparator): Single dose of 133 mg (10 mL) EXPAREL (bupivacaine liposome injectable suspension) expanded in volume with 10 mL of normal saline for a total volume of 20 mL.
  Interventions: Drug: bupivacaine liposome injectable suspension
- EXPAREL 266 mg (Active Comparator): Single dose of 266 mg (20 mL) EXPAREL (bupivacaine liposome injectable suspension).
  Interventions: Drug: bupivacaine liposome injectable suspension
- Placebo (Placebo Comparator): Normal saline (20 mL).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: bupivacaine liposome injectable suspension — bupivacaine liposome injectable suspension 133 mg expanded with normal saline to 20 mL or 266 mg in 20 mL
  Other Names: EXPAREL
  Arms: EXPAREL 133 mg; EXPAREL 266 mg
Drug: Placebo — Normal saline.
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
This is a Phase 3, multicenter, randomized, double-blind, placebo-controlled study in 232 adult subjects undergoing primary unilateral TKA under general or spinal anesthesia.

DETAILED DESCRIPTION:
On Day 0, eligible subjects will be randomized in a 1:1:1 ratio to receive a single dose of either EXPAREL 133 mg in 10 mL expanded in volume with 10 mL of normal saline for a total volume of 20 mL (Group 1); EXPAREL 266 mg in 20 mL (Group 2); or placebo 20 mL (Group 3). Study drug (EXPAREL or placebo) will be administered in a blinded manner via an ultrasound guided single-dose femoral nerve block at least 1 hour prior to surgery. Prior to placement of the prosthesis, 8 mL of bupivacaine hydrochloride (HCl) (0.5%) diluted with 8 mL of normal saline will be administered by the surgeon as a periarticular infiltration to the posterior capsule (8 mL medially and 8 mL laterally).

Postsurgical assessments will include pain intensity scores using a 10-cm visual analog scale (VAS); total postsurgical opioid consumption; overall benefit of analgesia score (OBAS) questionnaire; subject satisfaction with overall analgesia using a 5-point Likert scale; neurological assessment; sensory function assessment; motor function assessment; the study physical therapy assessments (ie, timed walk, timed up and go, and stair climbing tests); discharge readiness; unscheduled phone calls or office visits related to pain; 12-lead ECGs; vital sign measurements; and clinical laboratory tests. Adverse events will be recorded from the time the informed consent form (ICF) is signed through postsurgical Day 29.

Follow-up visits will be scheduled for all subjects on postsurgical Days 6 and 10. A follow-up phone call will be made on postsurgical Day 29.

Pharmacokinetic (PK) parameters will be estimated from plasma bupivacaine measurements using non-compartmental analysis based on the sampling schedule of baseline (prior to the nerve block) through postsurgical Day 10.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, at least 18 years of age at screening.
2. Scheduled to undergo primary unilateral TKA under general or spinal anesthesia.
3. American Society of Anesthesiologists (ASA) physical status 1, 2, or 3.
4. Female subject must be surgically sterile; or at least 2 years postmenopausal; or have a monogamous partner who is surgically sterile; or practicing double-barrier contraception; or practicing abstinence (must agree to use double-barrier contraception in the event of sexual activity); or using an insertable, injectable, transdermal, or combination oral contraceptive approved by the FDA for greater than 2 months prior to screening and commit to the use of an acceptable form of birth control for the duration of the study and for 30 days after completion of the study.
5. Able to demonstrate sensory function by exhibiting sensitivity to cold, pinprick, and light touch.
6. Able to provide informed consent, adhere to the study visit schedule, and complete all study assessments.

Exclusion Criteria:

1. Currently pregnant, nursing, or planning to become pregnant during the study or within 1 month after study drug administration.
2. Planned concurrent surgical procedure (e.g., bilateral TKA).
3. Concurrent painful physical condition that may require analgesic treatment (such as an NSAID or opioid) in the postsurgical period for pain that is not strictly related to the knee surgery and which may confound the postsurgical assessments (e.g., significant pain from other joints including the non-index knee joint, chronic neuropathic pain, concurrent or prior contralateral TKA, concurrent foot surgery).
4. Previous open knee surgery on the knee being considered for TKA. Prior arthroscopy is permitted.
5. History of hypersensitivity or idiosyncratic reaction to amide-type local anesthetics.
6. Contraindication to any one of the following: bupivacaine, oxycodone, morphine, or hydromorphone.
7. Use of any of the following medications within the times specified before surgery: long-acting opioid medication or NSAIDs (except for low-dose aspirin used for cardioprotection) within 3 days, or any opioid medication within 24 hours.
8. Initiation of treatment with any of the following medications within 1 month of study drug administration or if the medication(s) are being given to control pain: selective serotonin reuptake inhibitors (SSRIs), selective norepinephrine reuptake inhibitors (SNRIs), gabapentin, pregabalin (Lyrica®), or duloxetine (Cymbalta®). If a subject is taking one of these medications for a reason other than pain control, he or she must be on a stable dose for at least 1 month prior to study drug administration.
9. Current use of systemic glucocorticosteroids within 1 month of enrollment in this study.
10. Use of dexmedetomidine HCl (Precedex®) within 3 days of study drug administration.
11. History of impaired kidney function, poorly controlled chronic respiratory disease, rheumatoid arthritis, coagulopathy, or loss of sensation in extremities.
12. Impaired kidney function (e.g., serum creatinine level >2 mg/dL [176.8 µmol/L] or blood urea nitrogen level >50 mg/dL [17.9 mmol/L]) or impaired liver function (e.g., serum aspartate aminotransferase [AST] level >3 times the upper limit of normal [ULN] or serum alanine aminotransferase [ALT] level >3 times the ULN.)
13. Uncontrolled anxiety, psychiatric, or neurological disorder that might interfere with study assessments.
14. Any chronic neuromuscular deficit effecting the peripheral nerves or muscles of the surgical extremity.
15. Any chronic condition or disease that would compromise neurological or vascular assessments.
16. Malignancy in the last 2 years, with the exception of non-metastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix.
17. Suspected or known history of drug or alcohol abuse within the previous year.
18. Body weight <50 kg (110 pounds) or a body mass index >44 kg/m2.
19. Previous participation in an EXPAREL study.
20. Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2016-06-03; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James B Jones, MD, PharmD, Study Director — Pacira Pharmaceuticals, Inc
Locations (17):
- United States (14):
  - Horizon Research Group, Inc, Mobile, Alabama
  - Denver Metro Orthopedics, Englewood, Colorado
  - Jackson Memorial Hospital/University of Miami, Miami, Florida
  - Pensacola Research Associates, Pensacola, Florida
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Montefiore Medical Center, The Bronx, New York
  - Fairview Hospital, Cleveland, Ohio
  - Indiana Regional Medical Center, Indiana, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Chan Soon-Shiong Medical Center, Windber, Pennsylvania
  - Hermann Drive Surgical Hospital, Houston, Texas
  - Westside Surgical Hospital, Houston, Texas
  - Southampton Orthopaedics Sports Medicine, Franklin, Virginia
- Ziekenhuis Oost-Limburg, Genk, Belgium
- Denmark (2):
  - Aarhus University Hospital, Aarhus C
  - Regionshospital Silkeborg, Silkeborg

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between June 3, 2016 and June 30, 2017 at 13 sites in the US and Europe
Groups:
- EXPAREL 133 mg: 10 mL EXPAREL (bupivacaine liposome injectable suspension) expanded with 10 mL normal saline as single-injection femoral nerve block ≥1 h preoperatively
- EXPAREL 266 mg: 20 mL EXPAREL (bupivacaine liposome injectable suspension) as single-injection femoral nerve block ≥1 h preoperatively
- Placebo: 20 mL normal saline as single-injection femoral nerve block ≥1 h preoperatively
Period: Overall Study
Arm/Group | EXPAREL 133 mg | EXPAREL 266 mg | Placebo
Started | 76 | 77 | 79
Completed | 75 | 73 | 74
Not Completed | 1 | 4 | 5

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received study drug, with analysis by actual treatment received.
Groups:
- Total: Total of all reporting groups
Arm/Group | EXPAREL 133 mg | EXPAREL 266 mg | Placebo | Total
Number analyzed (Participants) | 75 | 76 | 79 | 230
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (6.94) | 66.0 (9.01) | 65.4 (8.69) | 65.3 (8.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 43 | 53 | 132
  Male | 39 | 33 | 26 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 2 | 6
  Not Hispanic or Latino | 73 | 74 | 75 | 222
  Unknown or Not Reported | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 5 | 12 | 25
  White | 66 | 69 | 67 | 202
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Belgium | 36 | 37 | 36 | 109
  United States | 38 | 38 | 40 | 116
  Denmark | 1 | 1 | 3 | 5
Visual analog scale pain score [Mean (Standard Deviation); unit: cm] — Visual Analog Scale (VAS) is a pain scale. The VAS was presented as a straight 10 cm line, where 0 cm is no pain and 10 cm is the worst pain possible. Patients were asked, "How much pain are you experiencing right now? Please place a vertical mark on the line below to indicate the level of pain you are experiencing right now."
  cm | 2.12 (2.656) | 2.08 (2.546) | 1.80 (2.195) | 1.99 (2.458)
American Society of Anesthesiologists classification [Count of Participants; unit: Participants] — American Society of Anesthesiologists (ASA) classification was determined by physicians using the ASA Physical Status Classification System which assesses the patient's pre-anesthesia medical co-morbidities. ASA 1 patients would be considered a normal, healthy patient. ASA 2 is a patient with mild systemic disease(eg, smoker, well controlled diabetes or high blood pressure (HBP)). ASA 3 is a patient with severe systemic disease (eg poorly controlled diabetes or HBP). ASA 4 is a patient with severe systemic disease that is a constant threat to life (eg, recent myocardial infarction, stroke).
  Participants
    Score: 1 | 11 | 9 | 10 | 30
    Score: 2 | 41 | 41 | 46 | 128
    Score: 3 | 23 | 26 | 23 | 72
    Score: Greater than or equal to 4 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of Visual Analog Scale (VAS) Pain Intensity Scores Through 72 Hours
Description: AUC of VAS pain intensity scores through 72 hours. Visual Analog Scale (VAS) is a pain scale. The VAS was presented as a straight 10 cm line, where 0 cm is no pain and 10 cm is the worst pain possible. Patients were asked, "How much pain are you experiencing right now? Please place a vertical mark on the line below to indicate the level of pain you are experiencing right now."
Time Frame: 0-72 hours
Population: Efficacy population: all participants who received study drug and underwent the surgery, with analysis based on randomized treatment
Measure: Least Squares Mean (Standard Error); unit: cm*hr
Arm/Group | EXPAREL 133 mg | EXPAREL 266 mg | Placebo
Number analyzed (Participants) | 75 | 76 | 79
cm*hr | 259.545 (19.011) | 250.998 (18.849) | 279.794 (18.493)
Statistical Analysis 1: Comparison: EXPAREL 133 mg vs Placebo; Test type: Superiority; p = 0.4463, ANOVA; LSMD = -20.249, 95% CI 2-sided [-72.361 to 31.864]
Statistical Analysis 2: Comparison: EXPAREL 266 mg vs Placebo; Test type: Superiority; p = 0.2749, ANOVA; LSMD = -28.796, 95% CI 2-sided [-80.483 to 22.892]

2. Secondary Outcome: Total Postsurgical Opioid Consumption Through 72 Hours
Description: Total postsurgical opioid consumption (converted to IV morphine equivalents) through 72 hours
Time Frame: 0-72 hours
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg
Arm/Group | EXPAREL 133 mg | EXPAREL 266 mg | Placebo
Number analyzed (Participants) | 75 | 76 | 79
mg | 69.466 (4.403) | 74.393 (4.669) | 81.469 (5.006)
Statistical Analysis 1: Comparison: EXPAREL 133 mg vs Placebo; Test type: Superiority; p = 0.0716, ANOVA; LSM treatment ratio = 0.853, 95% CI 2-sided [0.717 to 1.014]
Statistical Analysis 2: Comparison: EXPAREL 266 mg vs Placebo; Test type: Superiority; p = 0.3004, ANOVA; LSM treatment ratio = 0.913, 95% CI 2-sided [0.769 to 1.084]

3. Secondary Outcome: Percentage of Opioid-free Participants Through 72 Hours
Description: Percentage of participants who did not receive opioid medication through 72 hours
Time Frame: 0-72 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | EXPAREL 133 mg | EXPAREL 266 mg | Placebo
Number analyzed (Participants) | 75 | 76 | 79
Participants | 0 | 0 | 0

4. Secondary Outcome: Time to First Opioid Rescue Through 72 Hours
Description: Time to first opioid rescue medication consumed through 72 hours. The "time to rescue" is estimated for each quartile from the Kaplan-Meier analysis, in which first quartile represents the time it took for the first 25% of the population to receive rescue medication, median quartile represents the time it took 50% of the population to receive rescue medication, and third quartile represents the time it took 75% of the population to receive rescue medication.
Time Frame: 0-72 hours
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: h
Arm/Group | EXPAREL 133 mg | EXPAREL 266 mg | Placebo
Number analyzed (Participants) | 75 | 76 | 79
h
  First quartile | 1.80 [0.87 to 2.22] | 1.53 [0.75 to 2.13] | 1.08 [0.65 to 1.65]
  Second quartile | 3.03 [2.38 to 3.85] | 2.87 [2.25 to 3.47] | 2.40 [1.68 to 2.90]
  Third quartile | 5.07 [4.15 to 7.25] | 5.78 [3.98 to 8.12] | 3.72 [3.15 to 5.07]
Statistical Analysis 1: Comparison: EXPAREL 133 mg vs Placebo; The overall distribution as estimated by the Kaplan-Meier analysis was compared between the EXPAREL arm and the placebo arm; Test type: Superiority; p = 0.1896, Log Rank
Statistical Analysis 2: Comparison: EXPAREL 266 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.2549, Log Rank

ADVERSE EVENTS:
Time Frame: From screening to day 29 postsurgery
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans whether or not considered drug-related. An AE could therefore have been any unfavorable and unintended sign (eg, abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug without any judgment about causality. Serious AEs were defined as per clinicaltrials.gov.
Arm/Group | EXPAREL 133 mg | EXPAREL 266 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/76 | 0/79
Serious Adverse Events (participants affected / at risk) | 5/75 | 8/76 | 6/79
Other Adverse Events (participants affected / at risk) | 73/75 | 74/76 | 76/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EXPAREL 133 mg (N=75) | EXPAREL 266 mg (N=76) | Placebo (N=79)
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Sinus arrest (Cardiac disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0
Postprocedural hematoma (Injury, poisoning and procedural complications) | 3 | 1 | 0
Postprocedural swelling (Injury, poisoning and procedural complications) | 1 | 0 | 0
Motor dysfunction (Nervous system disorders) | 0 | 2 | 0
Transient ischemic attack (Nervous system disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EXPAREL 133 mg (N=75) | EXPAREL 266 mg (N=76) | Placebo (N=79)
Motor dysfunction (Nervous system disorders) | 34 | 35 | 34
Dizziness (Nervous system disorders) | 3 | 7 | 5
Dysgeusia (Nervous system disorders) | 3 | 2 | 6
Sensory loss (Nervous system disorders) | 2 | 6 | 1
Headache (Nervous system disorders) | 4 | 2 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 4
Nausea (Gastrointestinal disorders) | 27 | 34 | 24
Constipation (Gastrointestinal disorders) | 12 | 16 | 15
Vomiting (Gastrointestinal disorders) | 4 | 10 | 9
Dyspepsia (Gastrointestinal disorders) | 2 | 5 | 2
Pyrexia (General disorders) | 23 | 18 | 22
Peripheral swelling (General disorders) | 0 | 7 | 3
Muscle twitching (Musculoskeletal and connective tissue disorders) | 5 | 7 | 4
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 2 | 5
Hepatic enzyme increased (Investigations) | 7 | 1 | 3
Hemoglobin decreased (Investigations) | 1 | 3 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 8 | 10
Hypotension (Vascular disorders) | 8 | 4 | 5
Urinary retention (Renal and urinary disorders) | 3 | 10 | 8
Fall (Injury, poisoning and procedural complications) | 4 | 5 | 0
Postprocedural hematoma (Injury, poisoning and procedural complications) | 4 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 5 | 5 | 5
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0
Confusional state (Psychiatric disorders) | 1 | 2 | 4
Anemia (Blood and lymphatic system disorders) | 1 | 6 | 5
Insomnia (Psychiatric disorders) | 1 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results conducted at Site shall not be published before 1st multicenter publication by Sponsor but can proceed if there is no such publication ≤18 months after study completion/termination at all sites and all data have been received. Before submitting manuscript/materials to an outside person/entity, site shall give Sponsor 60 days to review and comment. Site shall, upon request, further delay publication/presentation for ≤120 days to allow Sponsor to protect its interests in Inventions.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-06-20): https://cdn.clinicaltrials.gov/large-docs/78/NCT02713178/SAP_000.pdf
  • Study Protocol (2016-11-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT02713178/Prot_001.pdf